CLINICAL TRIAL: NCT07405853
Title: A Randomised, Partly Blinded Investigation to Evaluate the Clinical Performance and Safety of pHyph in Adult Women With Vulvovaginal Candidiasis Compared With an Untreated Control Group
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gedea Biotech AB (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VVC-2025
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Vulvovaginal Candidiasis (VVC)
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pHyph treatment (Active Comparator): Application of vaginal tablet every day for 6 days
  Interventions: Device: pHyph
- No treatment (No Intervention)

INTERVENTIONS:
Device: pHyph — pHyph is a vaginal tablet lowering the vaginal pH
  Arms: pHyph treatment

SUMMARY:
The goal of this clinical trial is to learn if pHyph works to reduce signs and symptoms of vulvovaginal candidiasis (thrush). It will also learn about the safety of pHyph. The main questions it aims to answer are:

* Does pHyph reduce the signs and symptoms of vulvovaginal candidiasis after an initial 6 day daily treatment?
* Does an additional 6 day treatment course after the initial one further reduce signs and symptoms of vulvovaginal candidiasis?
* What medical problems do participants have when applying pHyph? Researchers will compare pHyph to no treatment Day 0 to Day 7 to see if pHyph reduces signs and symptoms of vulvovaginal candidiasis. For patients that received initial treatment, researchers will also compare the treatment outcome Day 7 to the treatment outcome after an additional treatment course of pHyph, Day 14.

Participants will:

* Apply pHyph every day for 6 days or receive no treatment and visit the clinic 7 days after the initial screening visit. Patients that received treatment will continue with pHyph every day for 6 days and patients that did not receive any treatment will receive standard of care for vulvovaginal candidiasis and leave the study.
* Patients that receive pHyph will visit the clinic Day 0 (screening), Day 7, and Day 14, and have a telephone call Day 25. Patients that do not receive pHyph will visit the clinic Day 0 (screening) and Day 7.
* Keep a diary of their symptoms and confirm that they have applied pHyph.

DETAILED DESCRIPTION:
1. Full title A randomized, partly blinded investigation to evaluate the clinical performance and safety of pHyph in adult women with vulvovaginal candidiasis compared with an untreated control group
2. Rationale Vulvovaginal candidiasis (VVC) is a vaginal yeast infection that can cause abnormal vaginal discharge and often itching, affecting up to 75% of all women. Several approved drugs are already available for VVC, but they are not always effective, which means that the infection can recur.

   Given the limitations of current treatment and prevention strategies for vulvovaginal infections, as well as the high frequency of women misdiagnosing themselves, there is a need for new over-the-counter (OTC) treatment options that can treat both VVC and bacterial vaginosis, are safe during pregnancy, and have a low risk of resistance development.

   The treatment investigated in this research study is a medical device in the form of a vaginal tablet called pHyph. pHyph contains - glucono-delta-lactone, a substance that occurs naturally in the body, as it is a temporary substance in the breakdown of common sugar. It is also an approved food additive. In pHyph, glucono-delta-lactone causes the acidity (pH value) in the vagina to decrease to normal. In a slightly acidic environment, yeast fungi do not cause VVC in the same extent and lactobacilli are also favored, which can also inhibit yeast fungi.

   The main aim of the study is to investigate the change in signs and symptoms of VVC after 6 days of treatment with pHyph compared to an untreated control group.
3. Objectives

Primary objective:

To evaluate the change in signs and symptoms of VVC after 6 days of treatment with pHyph compared to an untreated control group.

Secondary objectives:

1. To further investigate the difference in clinical performance after 6 days of daily treatment with pHyph compared to no treatment (untreated control).
2. To investigate the difference in the absence of fungus after 6 days of daily treatment with pHyph compared to no treatment (untreated control).
3. To investigate the difference in clinical performance and absence of fungus after 6 days of daily treatment with pHyph compared to longer daily treatment.
4. To investigate the safety after a total of 12 days of daily treatment with pHyph as assessed by adverse events.

Exploratory objectives:

To evaluate vaginal microbiome data after 6 days of daily treatment with pHyph compared to no treatment (untreated control group).

To evaluate vaginal microbiome data after 6 days of daily treatment with pHyph compared to longer daily treatment.

4. Primary outcome measure The change in vulvovaginal signs and symptoms scores on day 7 compared to day 0.

1. By examining for signs of oedema, erythema, or excoriation of the vaginal mucosa and asking the patient about symptoms of itching, burning, and irritation. Signs and symptoms are scored using a rating scale from 0 to 3, at days 0 and 7.

5. Secondary outcome measure

The study will compare changes during and after treatment at different time points (days 0, 7, 14, and 25). Among other things, the following will be looked at:

* Presence of vaginal yeast infection
* Number of reported side effects
* Proportion of patients who experience reduction in symptoms such as itching, burning and irritation
* Change in vaginal pH
* How easy and user-friendly the treatment is perceived according to patients' responses in an app Exploratory outcome measure To further evaluate vaginal microbiome data for day 0, day 7, day 14 and day 25.

  6. Study design The study will include 48 research subjects with Vulvovaginal candidiasis. The research subjects will be divided into 2 groups; 32 who will receive treatment with pHyph and 16 who will receive no treatment at all. After 36 research subjects have been to visit 2, an evaluation of the data will be made. Depending on the outcome, the study can either be terminated or continue to include up to a maximum of 96 additional research subjects.

All research subjects will make 2 visits over a period of approximately 7-9 days. Participants receiving pHyph will have an additional clinic visit and a follow-up telephone call over a period of approximately 22-28 days 7. Study population The study will include women who have menstruated but not yet reached menopause, are 18 years of age or older, and have symptoms of VVC, such as itching, burning, and irritation in the genital area. The diagnosis of VVC is defined as having the following criteria: white or creamy discharge, at least 2 of the following signs and/or symptoms: edema, erythema, excoriations, itching, burning, or irritation of the vaginal mucosa scored at least 2 on a 0-3 rating scale, and visible yeast forms under a microscope. Participants may be recruited through advertising campaigns, social media, and mailings, among other methods. Women with signs of other vaginal infections will not be able to participate in the study.

8. Interventions The study involves a maximum of 3 clinical visits and a follow-up telephone call over a period of approximately 25 days, for the treatment group. The untreated group will attend 2 clinic visits. Participants receiving active treatment with pHyph will insert the vaginal tablets themselves at home at bedtime using a CE marked applicator. Detailed instructions will be given at the first visit. At the two (non-treatment group) and three (treatment group) clinical visits on days 0, 7, and 14, a gynecological examination and samples will be taken. Between visits, participants will answer questions about VVC symptoms and treatment via a mobile app.

* Visit 1 (Inclusion visit): study information, consent, and pregnancy test. A gynecological examination and sampling for VVC control will be performed. Participants receiving treatment will receive an applicator and tablets for 6 days of treatment to use at home each evening.
* Visit 2 (Day 7): Gynecological examination and sampling to check for VVC. Participants will answer questions about health and menstruation. Participants who receive treatment will receive additional tablets for 6 days and answer questions about the product's ease of use. Participants who do not receive treatment will end the study after this visit.
* Visit 3 (Day 14): Gynecological examination and sampling for VVC control. Participants are asked to answer questions about health and menstruation and questions about the ease of use of the product.
* Visit 4 (Day 25): Follow-up call by telephone. Participants are asked to answer questions about health and menstruation. Sampling for VVC control is performed by the participants themselves at home. The samples are sent in envelopes by post to the laboratory and the clinic according to instructions.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the clinical investigation, and to comply with all clinical investigation requirements.
2. Adult, post-menarchal, pre-menopausal women aged 18 years or older.
3. Diagnosis of VVC, defined as:

   * Having a white or creamy vaginal discharge, and
   * at least two signs (erythema, oedema and excoriation) and/or symptoms (itching, burning irritation) of VVC scored as at least 2 = moderate on a scale of 0-3, and
   * potassium hydroxide (KOH) or saline preparation from the inflamed vaginal mucosa or secretions revealing yeast forms (hyphae or pseudohyphae) or budding yeasts upon microscopic analysis.
4. Negative urine pregnancy test at screening.
5. Willing to refrain from using any intravaginal products (e.g., contraceptive creams, gels, foams, sponges, sex toys, lubricants or tampons, etc.) until EOT for the active treatment group (Day 14) or EOI for the no treatment group (Day 7).
6. Willing to use condoms during any sexual intercourse with a male sexual partner until EOT for the active treatment group (Day 14) or EOI for the no treatment group (Day 7).
7. Willing to use a method of contraception, e.g., condoms, hormonal contraception (oral, injectable, implantable, intravaginal, or transdermal), IUD (if a copper IUD is used, it must be combined with a condom) or intrauterine hormone-releasing system (IUS), during any sexual intercourse that might result in pregnancy from Visit 1 (Day 0) until EOI (Day 25 for the active treatment group or Day 7 for the no treatment group) to prevent pregnancy.

Exclusion Criteria:

1. Patients with known or apparent signs of other infectious causes of vaginal infection and/or vaginitis (e.g., BV, Trichomonas vaginalis, Neisseria gonorrhoeae, Chlamydia trachomatis, herpes simplex virus or human papillomavirus) at screening.
2. History of or presence at screening (Day 0) of any other clinically significant disease or disorder, medical/surgical procedure, or trauma, which, in the opinion of the Investigator, may either put the patient at risk because of participation in the clinical investigation, or influence the results or the patient's ability to participate in the clinical investigation.
3. Anticipated menstruation during the first treatment period (Day 0 until Day 7). If a patient is menstruating on Day 0, or if menstruation is anticipated during Days 0 to 7, inclusion can be postponed to an additional visit at a later date when the menstrual bleeding is no longer heavy (light bleeding or brown discharge is acceptable).
4. Patients who are pregnant or breastfeeding.
5. Patients who are planning to conceive within the 25 days of the investigation.
6. Patients who were treated for VVC (both OTC and prescription therapies) within the 14 days preceding screening.
7. Patients who are currently receiving antifungal therapy unrelated to VVC or have received antifungal therapy within the 14 days preceding screening.
8. Patients who have used any pH-modifying vaginal products within the 14 days preceding screening.
9. Patients who have received an investigational drug in a clinical trial within 30 days prior to screening.
10. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, to any of the product components.
11. The Investigator considers the patient unlikely to comply with clinical investigation procedures, restrictions and requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The change in CVVS score on Day 7 compared to that on Day 0. | From enrollment to Day 7
  The primary endpoint is defined as the numerical change in the CVVS score on Day 7 compared to that on Day 0.
  Each of the of the 6 VVC signs (erythema, oedema and excoriation) and symptoms (itching, burning and irritation) will be scored using the scale below:
  * 0 = none (absent)
  * 1 = mild (slight)
  * 2 = moderate (definitely present)
  * 3 = severe (marked, intense)
  The CVVS score is the sum of the six individual scores for vulvovaginal signs and symptoms.

SECONDARY OUTCOMES:
The proportion of patients having a reduction in CVVS score | As applicable from enrollment to Day 14
  Each of the of the 6 VVC signs (erythema, oedema and excoriation) and symptoms (itching, burning and irritation) will be scored using the scale below: • 0 = none (absent) • 1 = mild (slight) • 2 = moderate (definitely present) • 3 = severe (marked, intense) The CVVS score is the sum of the six individual scores for vulvovaginal signs and symptoms.
The proportion of patients having a reduction in the sum of the three vulvovaginal symptom scores (itching, burning and irritation). | As applicable from enrollment to Day 25
  The score is from 0-3 where 0 = no symptoms and 3 = Severe symptoms
The sum of the three vulvovaginal symptom scores (itching, burning and irritation). | As applicable from enrollment until Day 25
  The score is from 0-3 where 0 = no symptoms and 3 = Severe symptoms
Individual vulvovaginal symptom scores (itching, burning and irritation). | As applicable from enrollment to Day 25
  The score is from 0-3 where 0 = no symptoms and 3 = Severe symptoms
Other vulvovaginal symptom scores, as self-reported by patients. | As applicable from enrollment to Day 25
  Other vulvovaginal symptoms are scored from 0-3 where 0 is no symptoms and 3 is severe symptoms
The proportion of clinically cured patients, defined as having a CVVS score ≤3. | As applicable from enrollment to Day 14
  Each of the of the 6 VVC signs (erythema, oedema and excoriation) and symptoms (itching, burning and irritation) will be scored using the scale below: • 0 = none (absent) • 1 = mild (slight) • 2 = moderate (definitely present) • 3 = severe (marked, intense) The CVVS score is the sum of the six individual scores for vulvovaginal signs and symptoms.
The proportion of patients showing an absence of fungal hyphae in the wet smear. | As applicable from enrollment to Day 14
The proportion of mycologically cured patients, defined as vaginal cultures negative for growth of fungal species. | As applicable from enrollment to Day 25
The proportion of patients having both clinical cure according to secondary endpoint no. 7 as well as mycological cure according to secondary endpoint no. 9. | As applicable from enrollment to Day 14
The proportion of patients having both clinical cure according to secondary endpoint no. 7 as well as mycologically confirmed fungus at screening. | As applicable from enrollment to Day 14
The proportion of patients having a CVVS score = 0, i.e., the absence of all signs and symptoms. | As applicable from enrollment to Day 14
  Each of the of the 6 VVC signs (erythema, oedema and excoriation) and symptoms (itching, burning and irritation) will be scored using the scale below: • 0 = none (absent) • 1 = mild (slight) • 2 = moderate (definitely present) • 3 = severe (marked, intense) The CVVS score is the sum of the six individual scores for vulvovaginal signs and symptoms.
The change in CVVS score, i.e., the primary endpoint parameter, for patients that received treatment on Day 7-12. | From enrollment to Day 14
  Each of the of the 6 VVC signs (erythema, oedema and excoriation) and symptoms (itching, burning and irritation) will be scored using the scale below: • 0 = none (absent) • 1 = mild (slight) • 2 = moderate (definitely present) • 3 = severe (marked, intense) The CVVS score is the sum of the six individual scores for vulvovaginal signs and symptoms.
Change in vaginal pH | As applicable from enrollment to Day 14
The occurrence of vaginal yeasts, assessed by analysis (qPCR) of the vaginal microbiome, i.e., qPCR count of fungal species. | As applicable from enrollment to Day 25
Reported treatment-emergent adverse events (TEAEs) and device deficiencies in the active treatment group. | From enrollment to Day 25
Usability, measured by patient questionnaire administered via mobile application on Day 14. | From enrollment to Day 14
  Dichotomous questions and a question regarding general regard of the product using a 10 point scale where 1 is Not satisfied and 10 is Very satisfied

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - CTC, Ebbe Park, Linköping
  - CTC Stockholm, Solna
  - CTC, Uppsala

IPD SHARING:
Plan to Share IPD: No